CLINICAL TRIAL: NCT00771719
Title: Open-Label Exploratory, Multiple-Dose Study of Ceftobiprole to Evaluate the Pharmacokinetics and Broncho-Alveolar Penetration in Adults With Ventilator-Associated Pneumonia
Brief Title: Open Label Pharmacokinetic in Adult Patients With Ventilator-Associated Pneumonia
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study closed due to lack of enrollment; challenging patient population.
Sponsor: Basilea Pharmaceutica (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR015304; NOS-1002 (Other: Basilea (Internal Reference))
Record Dates: First submitted 2008-10-09; First posted 2008-10-13 (Estimated); Last update posted 2012-07-30 (Estimated); Status verified 2012-07

CONDITIONS: Ventilator Associated Pneumonia
Keywords: VAP
MeSH Terms: conditions — Pneumonia, Ventilator-Associated | interventions — ceftobiprole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ceftobiprole (Experimental): Ceftobiprole, 1 G q8h as 4 hour infusions for 2 days
  Interventions: Drug: Ceftobiprole

INTERVENTIONS:
Drug: Ceftobiprole — Ceftobiprole, 1 G q8h as 4 hour infusions for 2 days

SUMMARY:
The purpose of this research study is to measure the levels of ceftobiprole in the blood, urine and tissues of the lungs during and after administration of four doses of ceftobiprole. Safety of the drug will also be evaluated.

DETAILED DESCRIPTION:
Patients will receive a intravenous dose of ceftobiprole infused over 4 hours. Multiple blood samples will be obtained to determine the concentration of Ceftobiprole in the blood. Bronchoalveolar lavage (BAL) samples will be collected to determine the concentration of ceftobiprole in the BAL fluid. The penetration of the drug into the lung will be calculated. Four 1000mg administered every 8 hours

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent
* Between 18 and 75 years of age inclusive
* VAP - 48 hours after onset of mechanical ventilation
* BMI 18 - 35 inclusive
* Albumin < 3.3 g/dL or clinical evidence of edema
* Negative Pregnancy test
* Expected survival of at least 7 days

Exclusion Criteria:

* Renal impairment (CrCl < 80 mL/min)
* Known drug allergy (including penicillin, cephalosporin, carbapenems, or other beta-lactams)
* History of seizures
* Sustained shock, unresponsive to sympathomimetics
* Conditions that may have jeopardized adherence to the protocol (NYHA Class 4 cardiac disease, >15% total body burn or significant third degree burn)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2008-10; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (to measure the levels of ceftobiprole in the blood and urine and tissues of the lungs) during dosing and 24 hours after last dose infused | 2 days

SECONDARY OUTCOMES:
Safety will be evaluated throughout the study. | Study Duration

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- See also: Open Label pharmacokinetic in Adult Patients with Ventilator-Associated Pneumonia — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=792&filename=CR015304_CSR.pdf